CLINICAL TRIAL: NCT02254018
Title: An Open Phase I Single Dose Escalation Study of Bivatuzumab Mertansine Administered Intravenously in Patients With Advanced Squamous Cell Carcinoma of the Head and Neck With Repeated Administration in Patients With Clinical Benefit
Brief Title: Single Dose Escalation Study of Bivatuzumab Mertansine in Patients With Advanced Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1191.2
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — bivatuzumab mertansine

ARMS (1):
- bivatuzumab mertansine (Experimental): single dose escalation
  Interventions: Drug: bivatuzumab mertansine

INTERVENTIONS:
Drug: bivatuzumab mertansine

SUMMARY:
maximum tolerated dose (MTD), safety, pharmacokinetics, efficacy of bivatuzumab mertansine

ELIGIBILITY:
Inclusion Criteria:

1. male and female patients aged 18 years or older
2. patients with histologically confirmed squamous cell carcinoma of the head and neck
3. patients with local and / or regional recurrent disease or distant metastases who are refractory to or not amenable to established treatments
4. measurable tumour deposits by one or more radiological techniques (MRI, CT)
5. life expectancy of at least 6 months
6. Eastern Cooperative Oncology Group (ECOG) performance score ≤ 2
7. patients must have given written informed consent (which must be consistent with International Conference of Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation)

Exclusion Criteria:

1. hypersensitivity to humanised or murine antibodies, immunoconjugates or the excipients of the trial drugs
2. known secondary malignancy requiring therapy
3. active infectious disease
4. brain metastases
5. neuropathy grade 2 or above (excluding pre-existing neuropathy of cranial nerves due to surgery, radiotherapy or tumour growth)
6. absolute neutrophil count less than 1,500/mm3
7. platelet count less than 100,000/mm3
8. bilirubin greater than 1.5 mg/dl (> 26 μmol/L, système internationale (SI) unit equivalent)
9. aspartate amino transferase (AST) and/or alanine amino transferase (ALT) greater than 3 times the upper limit of normal
10. serum creatinine greater than 1.5 mg/dl (> 132 μmol/L, SI unit equivalent)
11. concomitant non-oncological diseases which are considered relevant for the evaluation of the safety of the trial drug
12. chemo- or immunotherapy within the past three weeks prior to treatment with the trial drug or during the trial
13. radiotherapy to head and neck region within the past four weeks before inclusion or during the trial
14. men and women who are sexually active and unwilling to use a medically acceptable method of contraception
15. pregnancy or lactation
16. treatment with other investigational drugs or participation in another clinical trial within the past three weeks before start of therapy or concomitantly with this trial
17. patients unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2002-09-01 (Actual); Primary Completion 2005-02-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of bivatuzumab mertansine | up to day 21

SECONDARY OUTCOMES:
Number of patients with adverse events | up to day 21
  grading according to the common toxicity criteria (CTC)
Number of patients with clinically significant changes in laboratory parameters | up to day 21
Number of patients with clinically significant changes in vital signs | up to day 21
Tumor response | up to 1 year
  according to the response evaluation criteria in solid tumours (RECIST)
Concentration of bivatuzumab mertansine | up to day 21
Concentration of CD44v6 recognising IgG antibodies (anti-CD44v6-IgG) | up to day 21
Number of patients with development of human anti-human antibodies (HAHA) | up to day 21

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency